## **Protocol Summary**

Study Acronym/Protocol #: AAA 13-02

06 Dec 2017

NCT02528500

## **PROTOCOL SUMMARY**

| Study Title | Early Feasibility Assessment of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis in the Treatment of Type IV Thoracoabdominal Aortic Aneurysms Involving the Visceral Branch Vessels |
|---|---|
| Protocol Number | AAA 13-02 |
| Sponsor | W. L. Gore & Associates, Inc. Medical Products Division Telephone: 800-437-8181 |
| Study Design | This is a non-randomized, multicenter study designed to assess the initial feasibility of the GORE® EXCLUDER® Thoracoabdominal Branch Endoprosthesis (TAMBE Device) |
| Study Objective | Assess the initial safety of the TAMBE Device implantation procedure in the treatment of Aortic Aneurysms Involving the Visceral Branch Vessels |
| Study Rationale | This study is designed to provide evidence to support the use of the TAMBE Device as an option for endovascular treatment of patients with Type IV Thoracoabdominal Aortic Aneurysms. |
| Study Endpoints | Primary endpoint: Procedural Safety - Absence of the following events through 30 days post-procedure: • Death • Stroke • Myocardial Infarction • Bowel Ischemia • Paraplegia • Respiratory Failure • Renal Failure • Procedural Blood Loss ≥1000 mL Secondary endpoints: Technical Success - All of the following: • Successful access to the necessary arterial sites • Successful deployment of all required TAMBE Device components and any required accessory components • Patency of all required TAMBE Device components and any required accessory components on completion angiography • Absence of surgical conversion within 24 hours of initiation of the procedure |

| | <b>Device integrity -</b> Absence of the following events through one year of follow-up: |
|---|---|
| | Loss of functional patency in any branch component due to thrombus or mechanical failure of the branch components |
| | <ul> <li>Loss of functional patency in the main body component(s) due to<br/>thrombus or mechanical failure of the main body component(s)</li> </ul> |
| | <ul> <li>Separation of the branch components from the main body component(s)</li> </ul> |
| | <ul> <li>Separation of the main body component(s) from the accessory<br/>components (Distal Bifurcated Component and / or contralateral limb<br/>components)</li> </ul> |
| | Individual components of technical success |
| | Individual components of device integrity at one month, six months and one year follow-up |
| | Patency (Primary, Assisted Primary and Secondary) |
| | Absence of Type I and Type III endoleaks at one month follow-up |
| | <b>,</b> |
| Subject Population | Cubicate with There are belowing Annual Acutic Annual response level in a the Microsoft |
| | Subjects with Thoracoabdominal Aortic Aneurysms Involving the Visceral Branch Vessels |
| Number of Subjects Treated | 10 |
| Number of Sites | Six in the United States |
| Expected Time to Complete Enrollment | 18 Months |
| Schedule of Events | Assessments at Pre-treatment: |
| | CT of chest, abdomen and pelvis |
| | Physical exam |
| | Creatinine measurement |
| | Assessments at Treatment: |
| | Angiography |
| | Assessments at Hospital Discharge: |
| | Physical exam |
| | Creatinine measurement |
| | Abdominal ultrasound (optional) |
| | Assessments at Follow-up (One month, six months, and annually |
| | through 5 years): |
| | CT of chest, abdomen and pelvis (not required at hospital discharge) Lumber onice Series X ray (4 views) (appual follow up only)* |
| | <ul> <li>Lumbar spine series X-ray (4 views) (annual follow-up only)*</li> <li>Physical exam</li> </ul> |
| | Creatinine measurement |
| | Abdominal ultrasound (optional) |
| | *As enrollment is closed for this study, for all subjects that have completed their one |
| | year follow-up prior to this protocol amendment being implemented, subjects will be |

## $\mathsf{GORE}^{\circledast}$ <code>EXCLUDER\$</code> Thoracoabdominal Branch Endoprosthesis MD134357 AAA 13-02 Protocol Revision # 2 Doc Type SP

| | expected to have radiograph assessments at their next annual follow-up exam (i.e. two year follow-up) and annually thereafter. |
|---|---|
| Anticipated Total Study Duration | 7 years from initiation of enrollment |